CLINICAL TRIAL: NCT00347867
Title: Improvement of Utero-Placental Perfusion and Fetal Growth in IUGR and PET by Administration of Sildenafil Citrate in Pregnancy
Brief Title: Viagra for the Treatment of IUGR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Viagra.CTIL
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2006-07-04 (Estimated); Status verified 2006-06

CONDITIONS: IUGR
Keywords: IUGR; PET; Pregnancy; Viagra; Sildenafil citrate

INTERVENTIONS:
Drug: Viagra administration in IUGR/PET pregnancies

SUMMARY:
It has been suggested that Viagra (or other drugs that inhibit PDE-5, the enzyme that normally inhibits blood vessels' ability to expand) may have beneficial effects in hypertensive pregnancy and, possibly, preeclampsia.The benefits of Viagra were observed without any reduction in maternal blood pressure, thereby dissociating hypertension per se from the loss of NO (nitrous oxide) signaling in the uterine circulation.Following publications, suggesting that sildenafil citrate used as a therapeutic agent may improve myometrial perfusion in IUGR gestations by promoting myometrial small artery vasodilatation, decreasing peripheral resistance and increasing flow within the uteroplacental bed, we intend to administer this medication to parturients where intauterine growth restriction and pregnancy associated hypertension have been diagnosed in an attempt to induce vasodilatation and improved uteroplacental perfusion resulting in improved fetal growth.

DETAILED DESCRIPTION:
Each participant will receive, after informed consent a 25 mg tablet of Viagra [sildenafil citrate ]orally. The uteroplacental perfusion will be measured using transvaginal and transabdominal ultrasound Doppler velocimetry studies, before and after 2, 4, and 24 hours of Viagra ingestion. If no significant side effects are recorded, the protocol will be repeated , 48 hours after the first tablet ingestion, but using 50 mg Viagra.In cases of positive and encouraging results and if no serious side effects are detected we shall consider repeated administration of the lowest effcetive dose of viagra in an attempt to prevent prematurity and possibly reach term.our study will evaluate the effects of Viagra on uterine blood flow changes during pregnancy, and possible changes in other systems that contribute to normal fetal growth and development, in parallel to monitoring general and possible deleterious effects on the retina or other possible maternal or fetal organs.

ELIGIBILITY:
Inclusion Criteria:

* IUGR/PET/Pregnancy weeks 24-33.
* Informed consent.

Exclusion Criteria:

* Maternal cardiovascular morbidity.
* Usage of any vasodilator medication
* Smoking
* Diabetes

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2006-07

PRIMARY OUTCOMES:
Uteroplacental perfusion
Fetal growth
Maternal and fetal safety

CONTACTS AND LOCATIONS:
Overall Officials: Zeev Blumenfeld, MD, Principal Investigator — RAMBAM Health Care Campus, Technion
Locations (1):
- RAMBAM Health Care Campus, Haifa, Israel